CLINICAL TRIAL: NCT00691405
Title: A Double-blind, Randomized, Multicenter, Two-part Parallel-group, Dose-ranging Study of Twice-daily and Once-daily (R,R) Formoterol in the Treatment of Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Dose Ranging Study of Arformoterol Given Once Daily Compared to Arformoterol Given Twice Daily in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 091-026
Record Dates: First submitted 2008-06-02; First posted 2008-06-05 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: COPD
Keywords: Arformoterol; (R,R)-formoterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- A1 (Experimental): Arformoterol 5 mcg BID for 14 days
  Interventions: Drug: Arformoterol tartrate inhalation solution
- A2 (Experimental): Arformoterol 15 mcg BID for 14 days
  Interventions: Drug: Arformoterol tartrate inhalation solution
- A3 (Experimental): Arformoterol 25 mcg BID for 14 days
  Interventions: Drug: Arformoterol tartrate inhalation solution
- A4 (Placebo Comparator): Placebo inhalation solution BID for 14 days
  Interventions: Drug: Placebo
- B1 (Experimental): Arformoterol 15 mcg QD for 14 days
  Interventions: Drug: Arformoterol tartrate inhalation solution
- B2 (Experimental): Arformoterol 25 mcg QD for 14 days
  Interventions: Drug: Arformoterol tartrate inhalation solution
- B3 (Experimental): Arformoterol 50 mcg QD for 14 days
  Interventions: Drug: Arformoterol tartrate inhalation solution
- B4 (Placebo Comparator): Placebo inhalation solution QD for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Arformoterol tartrate inhalation solution — Arformoterol 5 mcg BID
  Other Names: (R,R)-formoterol; Brovana
  Arms: A1
Drug: Arformoterol tartrate inhalation solution — Arformoterol 15 mcg BID
  Other Names: (R,R)-formoterol; Brovana
  Arms: A2
Drug: Arformoterol tartrate inhalation solution — Arformoterol 25 mcg BID
  Other Names: (R,R)-formoterol; Brovana
  Arms: A3
Drug: Placebo — Placebo inhalation solution BID
  Arms: A4
Drug: Arformoterol tartrate inhalation solution — Arformoterol 15 mcg QD
  Other Names: (R,R)-formoterol; Brovana
  Arms: B1
Drug: Arformoterol tartrate inhalation solution — Arformoterol 25 mcg QD
  Other Names: (R,R)-formoterol; Brovana
  Arms: B2
Drug: Arformoterol tartrate inhalation solution — Arformoterol 50 mcg QD
  Other Names: (R,R)-formoterol; Brovana
  Arms: B3
Drug: Placebo — Placebo inhalation solution QD
  Arms: B4

SUMMARY:
A dose ranging study to evaluate the safety, tolerability and efficacy of arformoterol (given once or twice a day) in subjects with COPD.

DETAILED DESCRIPTION:
This study is a double-blind, repeat-dose, randomized, multicenter, two-part, parallel-group, dose-ranging study of arformoterol and placebo in the treatment of subjects with COPD. Approximately 215 subjects will be randomized in this study. Study participation will consist of a total of eight (8) study visits over approximately ten (10) weeks for each subject. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Subject may be male or female and must be aged greater than or equal to 35 years on the day the informed consent is signed.
* Female subject less than or equal to 65 years of age must have a serum pregnancy test conducted at study start and confirmed negative. Subjects of childbearing potential must be using an acceptable method of birth control and agree to continue its use throughout the study.
* In order to be considered not of childbearing potential female subjects must be:

  * documented surgically sterile (defined as status post-hysterectomy or bilateral tubal ligation) OR
  * postmenopausal
* Subject must have a primary diagnosis of COPD, which may include components of chronic bronchitis and/or emphysema. Diagnosis can be made during the screening process.
* Subject must have a minimum smoking history of 15 pack-years (pack-years = the number of cigarette packs per day times the number of years).
* Subject must have a chest x-ray that is consistent with the diagnosis of COPD (e.g., not diagnostic of pneumonia, other infection, atelectasis, or pneumothorax) and taken less than or equal to 6 months before study start. If there is no chest x-ray taken less than or equal to 6 months before study start, a chest x-ray will be performed at Visit 1.
* Subject must be able to complete all study questionnaires and logs reliably.

Exclusion Criteria:

* A female who is pregnant or lactating.
* Subject who has participated in an investigational drug study within 30 days prior to study start, or who is currently participating in another investigational drug study.
* Subject's schedule or travel prevents the completion of all required visits.
* Subject is scheduled for in-patient hospitalization, including elective surgery (in patient or out-patient) during the trial.
* Subject has had a life-threatening/unstable respiratory status, including upper or lower respiratory tract infection, within the 30 days prior to study start.
* Subject has a known history of asthma (except childhood asthma) or any chronic respiratory disease (including a current history of sleep apnea) other than COPD (chronic bronchitis and/or emphysema).
* Subject has a known history of alpha 1 antitrypsin deficiency-related emphysema.
* Subject has a history of cancer except non-melanoma skin cancer. Subjects with a history of cancer that is considered surgically cured and without a recurrence within the past 5 years may participate in the study. History of hematologic/lymphatic malignancy treated with chemotherapy or radiation is not allowed, under any condition.
* Subject has a history of lung resection of more than one full lobe or being a recipient of a lung or major organ transplant.
* Subject requires continuous supplemental oxygen therapy (unless subject resides at elevation greater than or equal to 4,000 feet).
* Subject has had a change in dose or type of any medications for COPD within 14 days before the screening visit.
* Subject has a known sensitivity to arformoterol, ipratropium or albuterol or any of the excipients contained in any of these formulations.
* Subject has a history of substance abuse within 12 months of Visit 1, or with a positive urine drug screen at study start.
* Subject is using any prescription drug for which concomitant beta-agonist administration is contraindicated (e.g., beta-blockers).
* Subject has had significant blood loss (>500 cc) or donated blood within 60 days preceding screening or plans to donate blood during or within 60 days after completing the study.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2003-10; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Part A: The primary efficacy endpoint is the time-normalized area under the FEV1 percent change from pre-dose curve over 12 hours (nAUC0-12) after the first (AM) dose at the 24 hour clinic visit (Visit 4) following 14 days of double-blind treatment. | Visit 2 (Day 0), Visit 3 (Day 7), Visit 4 (Day 14), Visit 5 (Day 21), Visit 6 (Day 28), Visit 7 (Day 42), Visit 8 (Day 48)
Part B: The primary efficacy endpoint is the time-normalized area under the FEV1 percent change from pre-dose curve over 24 hours (nAUC0-24) at the 24 hour clinic visit (Visit 7) following 14 days of double-blind treatment. | Visit 2 (Day 0), Visit 3 (Day 7), Visit 4 (Day 14), Visit 5 (Day 21), Visit 6 (Day 28), Visit 7 (Day 42), Visit 8 (Day 48)

SECONDARY OUTCOMES:
Relationship between plasma concentrations of arformoterol and changes in ECG QTc intervals at steady state throughout the dosing interval. | Visit 2 (Day 0), Visit 3 (Day 7), Visit 4 (Day 14), Visit 5 (Day 21), Visit 6 (Day 28), Visit 7 (Day 42), Visit 8 (Day 48)
Part A only: Time-normalized area under the curve for FEV1 percent change from pre-dose over 24 hours (nAUC0-24) for each 24 hour clinic visit. | Visit 2 (Day 0), Visit 3 (Day 7), Visit 4 (Day 14),
Part B only: Time-normalized area under curve for the FEV1 percent change from pre-dose over 12 hours (nAUC0-12) for each 24 hour clinic visit. | Visit 5 (Day 21), Visit 6 (Day 28), Visit 7 (Day 42), Visit 8 (Day 48)
Time-normalized area under the curve for the percent change in FEV1 from pre-dose over 6 hours (nAUC0-6) for the 6 hour clinic visit (Visits 3 and 6). | Visit 2 (Day 0), Visit 3 (Day 7), Visit 4 (Day 14), Visit 5 (Day 21), Visit 6 (Day 28), Visit 7 (Day 42), Visit 8 (Day 48)
Percent change in FEV1 from pre-dose to each post dose time point | Visit 2 (Day 0), Visit 3 (Day 7), Visit 4 (Day 14), Visit 5 (Day 21), Visit 6 (Day 28), Visit 7 (Day 42), Visit 8 (Day 48)
Peak percent change in FEV1 post-dose | Visit 2 (Day 0), Visit 3 (Day 7), Visit 4 (Day 14), Visit 5 (Day 21), Visit 6 (Day 28), Visit 7 (Day 42), Visit 8 (Day 48)
Ipratropium bromide metered-dose inhaler (MDI) use and racemic albuterol MDI use | Visit 2 (Day 0), Visit 3 (Day 7), Visit 4 (Day 14), Visit 5 (Day 21), Visit 6 (Day 28), Visit 7 (Day 42), Visit 8 (Day 48)
Morning and evening peak expiratory flow rate (PEFR) | Visit 2 (Day 0), Visit 3 (Day 7), Visit 4 (Day 14), Visit 5 (Day 21), Visit 6 (Day 28), Visit 7 (Day 42), Visit 8 (Day 48)
Exacerbations of COPD | Visit 2 (Day 0), Visit 3 (Day 7), Visit 4 (Day 14), Visit 5 (Day 21), Visit 6 (Day 28), Visit 7 (Day 42), Visit 8 (Day 48)
COPD symptom ratings | Visit 2 (Day 0), Visit 3 (Day 7), Visit 4 (Day 14), Visit 5 (Day 21), Visit 6 (Day 28), Visit 7 (Day 42), Visit 8 (Day 48)
Effects of withdrawal from therapy | Visit 2 (Day 0), Visit 3 (Day 7), Visit 4 (Day 14), Visit 5 (Day 21), Visit 6 (Day 28), Visit 7 (Day 42), Visit 8 (Day 48)
Relationship between plasma concentrations of (R,R)-formoterol and selected pharmacodynamic parameters. | Visit 2 (Day 0), Visit 3 (Day 7), Visit 4 (Day 14), Visit 5 (Day 21), Visit 6 (Day 28), Visit 7 (Day 42), Visit 8 (Day 48)
FEV1 percent change from pre-dose (24-hour trough) following 14 days of double-blind treatment. | Visit 2 (Day 0), Visit 3 (Day 7), Visit 4 (Day 14), Visit 5 (Day 21), Visit 6 (Day 28), Visit 7 (Day 42), Visit 8 (Day 48)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (31):
  - Encinitas, California
  - Long Beach, California
  - Brandon, Florida
  - Cleawater, Florida
  - Fort Lauderdale, Florida
  - Jacksonville, Florida
  - Port Orange, Florida
  - West Palm Beach, Florida
  - Austell, Georgia
  - Topeka, Kansas
  - Marrero, Louisiana
  - New Orleans, Louisiana
  - Opelousas, Louisiana
  - McCook, Nebraska
  - Princeton, New Jersey
  - Hickory, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Eugene, Oregon
  - Medford, Oregon
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Simpsonville, South Carolina
  - Spartanburg, South Carolina
  - Austin, Texas
  - San Antonio, Texas
  - Renton, Washington
  - Spokane, Washington
  - Tacoma, Washington